CLINICAL TRIAL: NCT06023199
Title: Assessing Functional Capacity in Sickle Cell Patients Receiving Voxelotor
Brief Title: Assessing Physical Function in Sickle Cell Patients Taking Voxelotor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U23-02-4988
Record Dates: First submitted 2023-08-07; First posted 2023-09-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voxeletor (Experimental)
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — Voxelotor is administered orally at a dose of 1500mg daily.
  Other Names: Oxbryta

SUMMARY:
Voxelotor is a novel hemoglobin polymerization inhibitor which has been demonstrated to reduce hemolysis and improve hemoglobin levels. There have been numerous studies examining the clinical impact of voxelotor in sickle cell disease (SCD) patients, but there are few published reports on the effects of treatment on physical function in patients with SCD. The hypothesis to be tested is that anemic SCD patients will have improvements in performance after 6 months of voxelotor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female,
4. aged 18-65 years
5. Diagnosis of sickle cell disease with HbSS, HbSc, HbS-beta thalassemia genotypes
6. Hemoglobin level of 6 g/dL - 10.5 g/dL
7. Between 0 and 10 vaso-occlusive (VOC) episodes in previous 12 months
8. Ability to take oral medication and be willing to adhere to the voxelotor regimen
9. For females of reproductive potential, they will be educated to avoid pregnancy during study period and for one month after due to limited data surrounding pregnancy and voxelotor
10. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
11. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Hemoglobin results < 6 g/dL or > 10.5 g/dL
2. Patients receiving hydroxyurea who have had a dose change within the prior 3 months
3. Females who are breastfeeding or pregnant
4. Patients who are receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) within 30 days of 6MWT
5. Any form of hepatic dysfunction as demonstrated by alanine aminotransferase (ALT) >4 × ULN or Child-Pugh Class C
6. Acute kidney injury or chronic renal disease with estimated glomerular filtration rate<30mL/min/1.73 m2
7. Current or previous diagnosis of malignancy within the last two years excluding local therapy for non-melanoma skin malignancy
8. Unstable cardiopulmonary disease within the last 6 months prior to study enrollment
9. Any conditions including behavioral or medical that in the opinion of the investigator, may negatively impact informed consent, participation and study interpretation
10. Current use of commercially available voxelotor
11. Prior hypersensitivity to voxelotor or its excipients
12. Patients with baseline gait and other physical impairments that would limit 6MWT and other functional assessment at discretion of the investigator
13. Patients who on day of assessment present with vaso-occlusive crisis or rate their pain greater than 6 on a scale of 1-10 using the Numeric Rating Scale will not be assessed that day and re-screened at the investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Participant's Physical Performance Using 6 Minutes Walk Test (6MWT) Pre and Post Treatment with Voxelotor. | 6 months from the treatment initiation
  The 6MWT is a sensitive objective assessment of functional exercise capacity which assess distance walked over 6 minutes.This test detects minor and moderate functional impairment resulting from treatment with Voxelotor.

OTHER OUTCOMES:
The Change in the Quality of Life as assessed by Sheehan Disability Scale (SDS) During the 6 Months Trial Period. | 6 months from the treatment initiation
  The SDS is a short self-reporting questionnaire that assess functional impairment in work/school, social and family life. The assessment scale has a total score of 30 (0 unimpaired and 30 extremely impaired).

CONTACTS AND LOCATIONS:
Overall Officials: Sheinei Alan, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenstaedt R, Penninx BW, Woodman RC. Anemia in the elderly: current understanding and emerging concepts. Blood Rev. 2006 Jul;20(4):213-26. doi: 10.1016/j.blre.2005.12.002. Epub 2006 Feb 10. PMID 16472893
- [Background] Vichinsky E, Hoppe CC, Ataga KI, Ware RE, Nduba V, El-Beshlawy A, Hassab H, Achebe MM, Alkindi S, Brown RC, Diuguid DL, Telfer P, Tsitsikas DA, Elghandour A, Gordeuk VR, Kanter J, Abboud MR, Lehrer-Graiwer J, Tonda M, Intondi A, Tong B, Howard J; HOPE Trial Investigators. A Phase 3 Randomized Trial of Voxelotor in Sickle Cell Disease. N Engl J Med. 2019 Aug 8;381(6):509-519. doi: 10.1056/NEJMoa1903212. Epub 2019 Jun 14. PMID 31199090
- [Background] Howard J, Ataga KI, Brown RC, Achebe M, Nduba V, El-Beshlawy A, Hassab H, Agodoa I, Tonda M, Gray S, Lehrer-Graiwer J, Vichinsky E. Voxelotor in adolescents and adults with sickle cell disease (HOPE): long-term follow-up results of an international, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Haematol. 2021 May;8(5):e323-e333. doi: 10.1016/S2352-3026(21)00059-4. Epub 2021 Apr 7. PMID 33838113
- [Background] Howard J, Hemmaway CJ, Telfer P, Layton DM, Porter J, Awogbade M, Mant T, Gretler DD, Dufu K, Hutchaleelaha A, Patel M, Siu V, Dixon S, Landsman N, Tonda M, Lehrer-Graiwer J. A phase 1/2 ascending dose study and open-label extension study of voxelotor in patients with sickle cell disease. Blood. 2019 Apr 25;133(17):1865-1875. doi: 10.1182/blood-2018-08-868893. Epub 2019 Jan 17. PMID 30655275
- [Background] Inusa BPD, Hsu LL, Kohli N, Patel A, Ominu-Evbota K, Anie KA, Atoyebi W. Sickle Cell Disease-Genetics, Pathophysiology, Clinical Presentation and Treatment. Int J Neonatal Screen. 2019 May 7;5(2):20. doi: 10.3390/ijns5020020. eCollection 2019 Jun. PMID 33072979
- [Background] Grosse SD, Odame I, Atrash HK, Amendah DD, Piel FB, Williams TN. Sickle cell disease in Africa: a neglected cause of early childhood mortality. Am J Prev Med. 2011 Dec;41(6 Suppl 4):S398-405. doi: 10.1016/j.amepre.2011.09.013. PMID 22099364
- [Background] Piel FB, Patil AP, Howes RE, Nyangiri OA, Gething PW, Dewi M, Temperley WH, Williams TN, Weatherall DJ, Hay SI. Global epidemiology of sickle haemoglobin in neonates: a contemporary geostatistical model-based map and population estimates. Lancet. 2013 Jan 12;381(9861):142-51. doi: 10.1016/S0140-6736(12)61229-X. Epub 2012 Oct 25. PMID 23103089
- [Background] Anie KA, Green J. Psychological therapies for sickle cell disease and pain. Cochrane Database Syst Rev. 2002;(2):CD001916. doi: 10.1002/14651858.CD001916. PMID 12076428
- [Background] Crawford J, Cella D, Cleeland CS, Cremieux PY, Demetri GD, Sarokhan BJ, Slavin MB, Glaspy JA. Relationship between changes in hemoglobin level and quality of life during chemotherapy in anemic cancer patients receiving epoetin alfa therapy. Cancer. 2002 Aug 15;95(4):888-95. doi: 10.1002/cncr.10763. PMID 12209734
- [Background] Corona LP, Andrade FCD, da Silva Alexandre T, de Brito TRP, Nunes DP, de Oliveira Duarte YA. Higher hemoglobin levels are associated with better physical performance among older adults without anemia: a longitudinal analysis. BMC Geriatr. 2022 Mar 21;22(1):233. doi: 10.1186/s12877-022-02937-4. PMID 35313814
- [Background] Yenamandra A, Marjoncu D. Voxelotor: A Hemoglobin S Polymerization Inhibitor for the Treatment of Sickle Cell Disease. J Adv Pract Oncol. 2020 Nov-Dec;11(8):873-877. doi: 10.6004/jadpro.2020.11.8.7. Epub 2020 Nov 1. PMID 33489427
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414